CLINICAL TRIAL: NCT03396393
Title: A Phase II, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Investigate the Safety, Pharmacokinetics and Efficacy of Dihydroartemisinin Tablets in Patients With Systemic Lupus Erythematosus
Brief Title: Exploratory Study of DHA in Systemic Lupus Erythematosus Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kunming Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY41078-201
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Dihydroartemisinin;Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — artenimol

STUDY DESIGN:
Intervention Model Description: Patients will be received DHA 40mg or DHA 80mg or DHA 120mg or placebo continuously for 24 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dihydroartemisinin 40mg (Experimental): Randomized 30 patients will be received Dihydroartemisinin tablets 40mg in oral continuously from Week 0 to Week 24 in addition to SOC.
  Interventions: Drug: Dihydroartemisinin tablet
- Dihydroartemisinin 80mg (Experimental): Randomized 30 patients will be received Dihydroartemisinin tablets 80mg in oral continuously from Week 0 to Week 24 in addition to SOC.
  Interventions: Drug: Dihydroartemisinin tablet
- Dihydroartemisinin 120mg (Experimental): Randomized 30 patients will be received Dihydroartemisinin tablets 120mg in oral continuously from Week 0 to Week 24 in addition to SOC.
  Interventions: Drug: Dihydroartemisinin tablet
- placebo (Placebo Comparator): Randomized 30 patients will be received placebo tablets in oral continuously from Week 0 to Week 24 in addition to SOC.
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Dihydroartemisinin tablet — DHA tablet
  Other Names: No other names
  Arms: Dihydroartemisinin 120mg; Dihydroartemisinin 40mg; Dihydroartemisinin 80mg
Drug: Placebo tablet — Placebo tablet
  Other Names: No other names
  Arms: placebo

SUMMARY:
The primary objective of the study is to assess the efficacy of DHA in patients with SLE.

DETAILED DESCRIPTION:
This is a Phase 2, multicentre, randomised, double-blind, placebo-controlled study to evaluate the Safety, Pharmacokinetics and Efficacy of four oral treatment regimens of DHA versus placebo while taking standard of care (SOC) treatment with corticosteroids in adult subjects with Systemic Lupus Erythematosus (SLE).

ELIGIBILITY:
Key Inclusion Criteria:

1. Fulfill at least 4 diagnostic criteria for SLE defined by American College of Rheumatology;
2. Positive antinuclear antibodies (ANA);
3. Activity Index (SLEDAI) score must be 6-11 points, inclusive;
4. Stable dose of prednisone (<30mg/d) for at least one month ;
5. Active mild to moderate SLE activity as demonstrated by British Isles Lupus Assessment Group Index (BILAG);
6. Males or females between 18 and 65 years old;
7. Weight of 45 kg or greater.

Key Exclusion Criteria:

1. Active Severe Lupus as defined by BILAG Index Level A or two or more of Level B in any body system/organ;
2. Subjects with concurrent relevant medical conditions like defined chronic infections or high risk of new significant infections;
3. Presence of active central nervous system (CNS) disease requiring treatment;
4. Subjects with active, severe SLE disease activity which involves the renal system;
5. Substance abuse or dependence;
6. History of malignant cancer within the last 5 years;
7. Subjects with any other condition which, in the investigator's judgment, would make the subject unsuitable for inclusion;
8. Subjects received any live vaccination within the 30 days prior to Visit 2;
9. Subjects received intravenous immunoglobulin (IVIg) or,plasmapheresis,or High dose prednisone or equivalent (> 100 mg/day) within 90 days prior to Visit 2;
10. Subjects who have had therapy with cyclophosphamide within 180 days prior to Visit 2 .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
SRI,Response at Week 24 according to a combined response index | week 24
  The combined response index incorporates the Bristish Isles Lupus Assessment Group (BILAG) assessment, the Systemic Lupus Eyrthematosus Disease Activity Index (SLEDAI), a physician's global assessment of disease activity, and treatment failure status.

SECONDARY OUTCOMES:
Change from baseline in SLEDAI score | week 4,8,12,16,20,24
  Change from baseline in SLEDAI score at week 4,8,12,16,20,24
Change from baseline in PAG score | week 4,8,12,16,20,24
  Change from baseline in PAG score at week 4,8,12,16,20,24
Number of days of daily prednisone dose Less than or equal to 7.5 mg/day | Baseline, Week 24
  Number of days of daily prednisone dose Less than or equal to 7.5 mg/day from baseline over 24 weeks
Percent of subjects with UPRO <0.5g/24h | Week 4,12,24
  Percent of subjects with UPRO <0.5g/24h from baseline at Week 4,12,24

CONTACTS AND LOCATIONS:
Overall Officials: Fengchun Zhang, Prof., Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: Undecided
This study has not been decided.